CLINICAL TRIAL: NCT00588965
Title: Effect of Beta-blocker Therapy on QTc Response in Exercise and Recovery in Normal Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MetroHealth Medical Center (Other)
Responsible Party: Principal Investigator, Elizabeth S. Kaufman, MD, Professor, Case Western Reserve University, MetroHealth Medical Center
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: IRB07-00418; NIH grant, GCRC MO1 RR000080
Record Dates: First submitted 2007-12-26; First posted 2008-01-09 (Estimated); Results first posted 2013-07-30 (Estimated); Last update posted 2013-07-30 (Estimated); Status verified 2013-07

CONDITIONS: Long QT Syndrome; Cardiac Repolarization
Keywords: QT interval; beta-blocker; exercise; electrocardiogram; repolarizaton
MeSH Terms: conditions — Long QT Syndrome; Motor Activity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Placebo Comparator): Subjects are assigned to placebo.
  Interventions: Drug: Placebo
- 2 (Active Comparator): Subjects will take propranolol LA 80 mg daily for one week then 160 mg for one week followed by the exercise test.
  Interventions: Drug: Propranolol LA

INTERVENTIONS:
Drug: Placebo — Placebo will be given 1 pill daily for a week, then 2 pills daily, followed by the exercise test.
  Arms: 1
Drug: Propranolol LA — Subjects will receive propranolol LA 80 mg one pill daily for 1 week then 2 pills daily for 1 week followed by exercise test.
  Arms: 2

SUMMARY:
Background. In congenital long QT syndrome type 1 (LQT1), episodes of ventricular tachycardia are usually triggered by exercise and can be prevented in most patients by beta-blocker therapy. In addition, LQT1 associated with a normal resting QT interval can be unmasked by the abnormal QT response to exercise testing (failure of the QT interval to shorten normally). Preliminary data from our laboratory show that the exercise QT intervals of patients with LQT1 are partially normalized by beta-blocker therapy. It is still currently not known if beta-blockers modify the QT/heart rate relationship (a primary effect on repolarization) or if the "normalizing" effect is due to the inability of subjects on beta-blockers to attain sufficiently high workloads (due to reduced heart rate) for prolongation to occur. Moreover, the physiologic response of the exercise QT interval to beta-blockers in healthy control subjects is not known.

Objective. The objective of this study is to define the impact of beta-blocker therapy on the QT response to exercise and recovery in normal subjects.

Methods. Approximately 36 healthy adult subjects age-matched to previously studied LQT1 subjects will undergo 1) screening history, 2) two weeks of beta-blocker therapy ending in an exercise test, and 3) two weeks of placebo therapy ending in an exercise test. Beta blocker and placebo will be given in random order in a double-blind fashion. The QT response to exercise and recovery will be compared between drug-free and beta-blocker-treated states. These data will be compared to those previously collected for LQT1 subjects.

Implications. These results will provide new information about the effect of beta-blocker therapy on repolarization parameters in normal subjects, and will provide a context in which to interpret the previous findings that beta-blocker administration modifies the QT response to exercise in LQT1 subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy normal adults, age- and gender-matched to previously studied LQT1 subjects

Exclusion Criteria:

* Cardiac disease
* Diabetes
* Hypertension
* Severe allergic reaction
* Asthma requiring treatment
* Use of medications other than oral contraceptives, acetaminophen, nonsteroidal anti-inflammatory drugs, or synthroid or other thyroid medications
* Pregnancy (subjects will be asked if they are pregnant)
* Inability to sign informed consent

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2007-08; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth S Kaufman, MD, Principal Investigator — MetroHealth Medical Center

RESULTS

PARTICIPANT FLOW:
Groups:
- All Participants: All participants were randomized to one of 2 sequences, in which they received either propranolol first, then placebo, or placebo first, then propranolol.
Period: Overall Study
Arm/Group | All Participants
Started | 35
Completed | 35
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- All Subjects: Subjects will take propranolol LA 80 mg or placebo daily for one week then propranolol LA 160 mg for one week or 2 placebo pills, followed by the exercise test. The participants will be randomized to one of 2 sequences: placebo first or propranolol first.
Arm/Group | All Subjects
Number analyzed (Participants) | 35
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 35
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 32 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 15
Region of Enrollment [Number; unit: participants]
  United States | 35

OUTCOME MEASURES:

1. Primary Outcome: QTc Response to Exercise on Versus Off Beta-blocker.
Description: To minimize the effect of heart rate on QT, QT was measured at heart rates between 100 and 110 beats per minute during exercise (on and off beta-blocker) and during recovery (on and off beta-blocker).
Time Frame: 2 weeks on each treatment then exercise test
Population: Please note that this was a crossover study. There were 35 subjects and each subject completed both the placebo and beta-blocker arm.
Measure: Mean (Standard Deviation); unit: ms
Arm/Group | Placebo | Propranolol
Number analyzed (Participants) | 35 | 35
ms
  During exercise | 320 (17) | 317 (16)
  During recovery | 317 (13) | 315 (14)

2. Secondary Outcome: Tpeak-end Interval (Tpe)
Description: Tpeak-end interval was measured at rest, exercise, and recovery on placebo and on propranolol.
Time Frame: Measured after 2 weeks on each intervention
Measure: Mean (Standard Deviation); unit: ms
Arm/Group | Placebo | Propranolol
Number analyzed (Participants) | 35 | 35
ms
  Rest | 74 (13) | 72 (13)
  Peak Exercise | 69 (13) | 61 (11)
  Recovery | 77 (19) | 68 (14)

ADVERSE EVENTS:
Groups:
- Placebo: Subjects are assigned to placebo.
- Propranolol: Subjects will take propranolol LA 80 mg daily for one week then 160 mg for one week followed by the exercise test.
Arm/Group | Placebo | Propranolol
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/35
Other Adverse Events (participants affected / at risk) | 0/35 | 0/35

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No